CLINICAL TRIAL: NCT03996785
Title: Investigations of Immediate and Short-term Effects of Nature Walks on Stress and Depression-related Symptoms
Brief Title: Effectiveness of Nature Walks in Depressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Marie-Claude Geoffroy, Assistant professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUSMD-18-33
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Experimental
Keywords: Clinical depression; Stress; Group-walking; Walking condition (nature vs urban)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were unaware as to whether they were assigned to an urban or nature walking condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban (Active Comparator): Patients will go for a silent 60-minute walk in an urban setting. The walk will take place in the months of June, July, August and September between 10:00 to 11:00 am.
  Participants will walk in groups of two to three participants accompanied by two research assistants trained in mental health (doctoral students in psychology). The urban walk will be located on Boulevard de la Vérendrye with large arteries with three to four lanes.
  Interventions: Behavioral: Walking in Urban setting
- Nature (Experimental): Patients will go for a silent 60-minute walk in a nature park setting. The walk will take place in the months of June, July, August and September between 10:00 to 11:00 am.
  Participants will walk in groups of two to three participants accompanied by two research assistants trained in mental health (doctoral students in psychology).
  The nature walk will take place at Parc Angrignon, an area of 96 hectares, one of Montreal's largest green and biodiverse spaces with a forest of 20 000 trees and a pond surrounded by willow trees.
  Interventions: Behavioral: Walking in nature setting

INTERVENTIONS:
Behavioral: Walking in Urban setting — Walking for 60 minutes as described above
  Arms: Urban
Behavioral: Walking in nature setting — Walking for 60 minutes as described above
  Arms: Nature

SUMMARY:
Over the past few years, a growing number of campaigns from around the world, including Canada, are highlighting the positive impact of spending time in nature on well-¬being. Indeed, mounting evidence suggests that spending time with nature is associated with a myriad of affective and cognitive benefits. Surprisingly few studies to date have tested the assumption that walking in nature versus in urban settings could alleviate stress and depressive symptoms in clinically depressed adults.

The main purpose of this study is to investigate the effectiveness of walking in nature versus in urban settings to improve depression related symptoms and reduce stress. The trial initially included 2 primary outcomes: patients stress levels (salivary cortisol) and depression-related symptoms (eg, affect, rumination, executive functioning).

However, due to hygienic concerns in light of the COVID-19 pandemic in 2020, the collection of saliva samples (and in turn, the measurement of stress levels via salivary cortisol) was removed from the study's procedure. The main outcome was changed to effects on positive and negative affect.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65 years, inclusively;
* Ability to speak French or English;
* Diagnosis major depressive disorder (DSM-IV);

Exclusion Criteria:

* Acute psychotic symptoms;
* Acute suicidal intent (within 48 hours);
* Unable to walk for 60 min or serious medical reasons (e.g. major surgery)
* Heart condition as per history or detected on electrocardiogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Change in affect from baseline up to 48 hours post-walk | Day 1 to Day 3
  Positive and Negative Affect Schedule (PANAS)

SECONDARY OUTCOMES:
Change in Executive Functions | The Stroop test will be administered at 2 time points: 1) before the walk (between 9:45-10:30); 2) after the walk (between 11:30-11:50)
  The stroop color word test is a widely used task to assess selective attention and inhibitory control. In the first block of this task (A), color words (red, blue, yellow, green) printed in black ink are presented in random order and participants are asked to read out loud the words. In the second block (B), solid color patches in one of the same four colors are shown and participants name the colors. Finally, in the third block (C), color words are printed in an incongruous ink color and participants must name the ink color (e.g. GREEN [typed in red]; response = red). Participants are asked to complete each block as quickly and accurately as possible and the time to complete each trial is calculated and averaged for each block. An interference score is calculated as followed: C - [(A + B) /2].
Change in suicidal Ideations | Day 1
  Severity of Suicidal Ideations The severity of current suicidal ideation will be assessed with three items derived from a prior study of momentary assessment of suicidal risk: "How intense is your desire to kill yourself right now"?; "How strong is your intention to kill yourself right now"?; "How strong is your ability to resist the urge to kill yourself right now"? Each item is scored on a scale from 0 (not strong [intense] at all) to 4 (very strong [intense]).
Change in depressive symptoms | Day 1 to Day 2
  The Beck Depression Inventory (BDI-II) The BDI is a widely used 21-item depression inventory with good internal consistency (α = .93 in the current sample) and validity. Items are answered on a 4-point scale from 0 to 3.
Change in rumination | Day 1
  The Rumination-Reflection Questionnaire (RRQ) The RRQ is a 24-item self-reported questionnaire assessing both self-rumination and self-reflection, 57 with 12 items corresponding to each subscale. Participants rate the degree to which they engage in self- rumination (e.g. "sometimes it is hard for me to shut off thoughts about myself") and self-reflective thoughts (e.g. "I love to meditate on the nature and meaning of things") on a Likert scale ranging from one (strongly disagree) to five (strongly agree)
Change in irritability | Day 1 to Day 3
  The Brief Irritability Test (BITe): The BITe is a 5-item self-report measure of irritability that is suitable for use among men and women. Participants respond to statements using a 6-point Likert scale ranging from Never to Always. Items include the following five statements: "I have been grumpy"; "I have been feeling like I might snap"; "Other people have been getting on my nerves".

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Geoffroy, PhD, Principal Investigator — McGill University
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No